CLINICAL TRIAL: NCT01013077
Title: The Effect of a New Emulsion in Dry Eye Patients on Tear Layer Aberrometry, Contrast Sensitivity, and Reading Ability.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern California College of Optometry at Marshall B. Ketchum University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, William Ridder, Professor, Southern California College of Optometry at Marshall B. Ketchum University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 09-11
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Dry Eye Syndrome
Keywords: functional vision; contrast sensitivity; aberrometry; reading ability
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Optive, Soothe, New Emulsion (Experimental): Subjects do not use artificial tears for one week followed by 1 month using Optive two times per day. One week washout then 1 month Soothe two times per day followed by one week washout and one month New Emulsion 2 times per day.
  Interventions: Other: Optive, Soothe, New Emulsion
- Soothe, New Emulsion, Optive (Experimental): Subjects do not use artificial tears for one week followed by 1 month using Soothe two times per day. One week washout then 1 month New Emulsion two times per day followed by one week washout and one month Optive 2 times per day.
  Interventions: Other: Soothe, New Emulsion, Optive
- New Emulsion, Optive, Soothe (Experimental): Subjects do not use artificial tears for one week followed by 1 month using New Emulsion two times per day. One week washout then 1 month Optive two times per day followed by one week washout and one month Soothe 2 times per day.
  Interventions: Other: New Emulsion, Optive, Soothe

INTERVENTIONS:
Other: Optive, Soothe, New Emulsion — One week without artificial tear use followed by Optive use a minimum of 2 drops per day for 1 month. One week without artificial tear use followed by Soothe use a minimum of 2 drops per day for 1 month. One week without artificial tear use followed by the New Emulsion use a minimum of 2 drops per day for 1 month.
  Arms: Optive, Soothe, New Emulsion
Other: Soothe, New Emulsion, Optive — One week without artificial tear use followed by Soothe use a minimum of 2 drops per day for 1 month. One week without artificial tear use followed by New Emulsion use a minimum of 2 drops per day for 1 month. One week without artificial tear use followed by the Optive use a minimum of 2 drops per day for 1 month.
  Arms: Soothe, New Emulsion, Optive
Other: New Emulsion, Optive, Soothe — One week without artificial tear use followed by New Emulsion use a minimum of 2 drops per day for 1 month. One week without artificial tear use followed by Optive use a minimum of 2 drops per day for 1 month. One week without artificial tear use followed by the Soothe use a minimum of 2 drops per day for 1 month.
  Arms: New Emulsion, Optive, Soothe

SUMMARY:
The purpose of this study is to investigate how the addition of a new emulsion artificial tear to the tear layer of dry eye and normal patients affects aberrometry, contrast sensitivity, and reading ability over time. Previous studies have indicated that daily use of artificial tears over a two week period decreases the short term affect of drop application on aberrometry and contrast sensitivity measurements. The present study will examine the effects of 4 weeks of artificial tear use to determine when the responses stabilize.

DETAILED DESCRIPTION:
Dry eye patients experience symptoms such as; irritation, dryness, a scratchy sensation, and blur. These symptoms are the result of an insufficient tear layer. Blur can occur in dry eye patients because of an irregular tear film surface.

Artificial tears are applied to the eye to treat a variety of eye conditions. These conditions typically are associated with dry eyes and include tear film deficiency due to ocular or systemic disease, lid resurfacing problems, and contact lens wear. The artificial tears are used to alleviate the dry eye symptoms.

Dry eye is a frequently encountered ocular condition. Recent studies estimate that 7.8% of women and 4.8% of men over the age of 50 suffer from dry eye. The administration of an artificial tear to the eye can disrupt the tear layer and this disruption could then result in a change in contrast sensitivity for a few moments. Aberrometry is a technique that is able to monitor tear layer disruption and its results may correlate with contrast sensitivity changes.

Tear layer disruption results in a decrease in the modulation transfer function (MTF) for the eye. Since the tear layer is the first refracting surface of the eye, its disruption can also result in a change in contrast sensitivity, visual acuity, and aberrometry. Previous work has demonstrated that higher order aberrations increase 1.44 fold after the tear film breaks up in normal subjects. Dry eye subjects demonstrate a significant increase in higher order aberrations (i.e., total S3+4+5, spherical-like S4, and coma-like S3+5) when compared to normal subjects. This has been interpreted to be the result of increased tear irregularities in the dry eye subjects.

When an artificial tear (i.e., Vismed) was applied to the tear layer of dry eye subjects, the optical aberrations decreased. This previous study only examined the short term affect (less than 10 minutes) of a single administration of an artificial tear. In this study, we propose to examine the short and long term effects of a new emulsion on contrast sensitivity, optical aberrations, and reading ability after administration into the tear layer of normal and dry eye subjects.

ELIGIBILITY:
Inclusion Criteria:

* mild, moderate, or severe symptoms of dry eye

Exclusion Criteria:

* uncontrolled systemic disease
* contact lens wear
* participation in another clinical trial
* best corrected visual acuity poorer than 20/25

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William H. Ridder, OD, PhD, Principal Investigator — Southern California College of Optometry at Marshall B. Ketchum University
Locations (1):
- Southern California College of Optometry, Fullerton, California, United States

IPD SHARING:
Plan to Share IPD: No
All data is available upon request.

REFERENCES:
- [Background] Thai LC, Tomlinson A, Ridder WH. Contact lens drying and visual performance: the vision cycle with contact lenses. Optom Vis Sci. 2002 Jun;79(6):381-8. doi: 10.1097/00006324-200206000-00012. PMID 12086305
- [Background] Ridder WH 3rd, Lamotte JO, Ngo L, Fermin J. Short-term effects of artificial tears on visual performance in normal subjects. Optom Vis Sci. 2005 May;82(5):370-377. doi: 10.1097/01.OPX.0000162646.30666.E3. PMID 15894913
- [Background] Ridder WH 3rd, LaMotte J, Hall JQ Jr, Sinn R, Nguyen AL, Abufarie L. Contrast sensitivity and tear layer aberrometry in dry eye patients. Optom Vis Sci. 2009 Sep;86(9):E1059-68. doi: 10.1097/OPX.0b013e3181b599bf. PMID 19648840

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the patients and staff of the clinic. The recruitment period was from 10/1/2009 till 7/30/2010.
Pre-assignment Details: The subjects were not allowed to use artificial tears for 1 week before the study started.
Groups:
- Optive, Soothe, New Emulsion: Optive was the first drop used followed by Soothe and then the New Emulsion.
- Soothe, New Emulsion, Optive: Soothe was the first drop used followed by the New Emulsion and then Optive.
- New Emulsion, Optive, Soothe: The New Emulsion was the first drop used followed by Optive and then Soothe..
Period: Overall Study
Arm/Group | Optive, Soothe, New Emulsion | Soothe, New Emulsion, Optive | New Emulsion, Optive, Soothe
Started | 7 | 7 | 6
Completed | 7 | 7 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The data from each drop was combined for all arms.
Groups:
- Optive, Soothe, New Emulsion: Drop order was Optive, then Soothe, then New Emulsion.
- Soothe, New Emulsion, Optive: Drop order was Soothe, then New Emulsion, then Optive.
- New Emulsion, Optive, Soothe: Drop order was New Emulsion, then Optive, then Soothe.
- Total: Total of all reporting groups
Arm/Group | Optive, Soothe, New Emulsion | Soothe, New Emulsion, Optive | New Emulsion, Optive, Soothe | Total
Number analyzed (Participants) | 7 | 7 | 6 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 6 | 20
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.8 (1.60) | 22.6 (1.67) | 24.4 (2.07) | 23.6 (1.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 4 | 17
  Male | 0 | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Contrast Sensitivity
Description: Change in contrast sensitivity with administration of the artificial tear. During a visit, contrast sensitivity is initially monitored for several minutes (i.e., pre-artificial tear application contrast sensitivity) and the artificial tear is then applied and the contrast sensitivity is continually measured for several more minutes (post-artificial tear application contrast sensitivity). The administration of the artificial tear decreases contrast sensitivity for approximately a minute. The data reported in the table is the change in contrast sensitivity from pre-artificial tear administration to the peak loss in contrast sensitivity after the artificial tear administration (negative values). This procedure is carried out before the subjects use artificial tears on a daily basis (i.e., baseline data) and for several weeks after using artificial tears on a daily basis (i.e., weeks 1, 2, and 4) to determine if there is an adaptation to the artificial tear.
Time Frame: Baseline, 1 week, 2 weeks, 4 weeks
Measure: Mean (Standard Error); unit: arbitrary units
Groups:
- Optive Normal; Soothe Normal: Commercial drop. Normal subjects.
- New Emulsion Normal: New formulation. Normal subjects.
- Optive Dry Eye; Soothe Dry Eye: Commercial drop. Dry eye subjects.
- New Emulsion Dry Eye: New formulation. Dry eye subjects.
Arm/Group | Optive Normal | Soothe Normal | New Emulsion Normal | Optive Dry Eye | Soothe Dry Eye | New Emulsion Dry Eye
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
arbitrary units
  Baseline | -0.375 (0.139) | -0.169 (0.133) | -0.313 (0.094) | -0.264 (0.117) | -0.268 (0.081) | -0.364 (0.063)
  Week 1 | -0.373 (0.111) | -0.118 (0.148) | -0.290 (0.081) | -0.275 (0.083) | -0.289 (0.113) | -0.446 (0.090)
  Week 2 | -0.186 (0.109) | -0.232 (0.138) | -0.178 (0.139) | -0.156 (0.076) | -0.226 (0.057) | -0.308 (0.109)
  Week 4 | -0.246 (0.123) | -0.366 (0.144) | -0.098 (0.074) | -0.433 (0.079) | -0.193 (0.051) | -0.386 (0.135)

ADVERSE EVENTS:
Groups:
- Optive; Soothe: Commercial drop.
- New Emulsion: New formulation.
Arm/Group | Optive | Soothe | New Emulsion
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days